CLINICAL TRIAL: NCT05065619
Title: A Phase I/II, Randomized, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of MT-2766 in Japanese Adults (COVID-19)
Brief Title: Safety Immunogenicity Study of MT-2766 in Japanese Adults（COVID-19）
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Public vaccination of approved ancestral strain COVID-19 vaccines will be terminated soon. And boosters must be dosed after ancestral vaccination approved in Japan. The study was terminated for ethical reason to prioritize the ancestral vaccination.
Sponsor: Medicago (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MT-2766-A-101/CP-PRO-CoVLP-028; jRCT2051210093 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2021-10-01; First posted 2021-10-04 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — MT-2766 vaccine; AS03 adjuvant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: MT-2766 High dose group and placebo group are randomized and observer-blinded. MT-2766 Low dose group is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MT-2766 High dose (3.75 µg) (Experimental)
  Interventions: Biological: MT-2766 High dose (3.75 µg)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MT-2766 Low dose (Experimental)
  Interventions: Biological: MT-2766 Low dose

INTERVENTIONS:
Biological: MT-2766 High dose (3.75 µg) — Subjects will receive two doses of MT-2766 high dose (3.75 µg) given 21 days apart into the deltoid region of the alternating arm (each arm will be injected once)
  Other Names: CoVLP, AS03 adjuvant
  Arms: MT-2766 High dose (3.75 µg)
Drug: Placebo — Subjects will receive two doses of placebo given 21 days apart into the deltoid region of the alternating arm (each arm will be injected once)
  Arms: Placebo
Biological: MT-2766 Low dose — Subjects will receive two doses of MT-2766 low dose given 21 days apart into the deltoid region of the alternating arm (each arm will be injected once)
  Other Names: CoVLP, AS03 adjuvant
  Arms: MT-2766 Low dose

SUMMARY:
The objective of this study is to evaluate the safety and immunogenicity of MT-2766 in Japanese adults.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must meet all of the following inclusion criteria at the Screening visit (Visit 1) and/or 1st vaccination visit (Visit 2) to be eligible for participation in this study. All Investigator assessment-based judgments must be carefully and fully documented in the source documents:

1. Subjects must have read, understood, and signed the informed consent form (ICF) prior to participating in the study; subjects must also complete study-related procedures and must communicate with the study staff at visits and by phone during the study;
2. At the Screening visit (Visit 1), Japanese male and female subjects must be ≥20 years of age;
3. At the Screening visit (Visit 1) and 1st vaccination visit (Visit 2), subject must have a body mass index (BMI) of ≥18.5 kg/m^2 and <30 kg/m^2;
4. Subjects are considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study;
5. Female subjects of childbearing potential must have a negative serum pregnancy test result at the Screening visit (Visit 1) and a negative urine pregnancy test result at 1st vaccination visit (Visit 2):

   Non-childbearing females are defined as:
   * Surgically sterile (defined as bilateral tubal ligation, hysterectomy or bilateral oophorectomy performed more than one month prior to the first study vaccination); OR
   * Post-menopausal (absence of menses for 12 consecutive months and age consistent with natural cessation of ovulation);
6. Female subjects of childbearing potential must use an effective method of contraception for one month prior to 1st vaccination visit (Visit 2) and agree to continue employing highly effective birth control measures for at least one month after the last study vaccination (or in the case of early termination, she must not plan to become pregnant for at least one month after her last study vaccination);
7. Subjects must be non-institutionalized (e.g. not living in rehabilitation centers or old-age homes);
8. Subjects have no acute or evolving medical problems prior to study participation and no clinically relevant abnormalities that could jeopardize subject safety or interfere with study assessments, as assessed by the Principal Investigator or sub-Investigator (thereafter referred as Investigator) and determined by medical history, physical examination, serology, clinical chemistry and hematology tests, urinalysis, and vital signs. Investigator discretion is permitted with this inclusion criterion.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria at the Screening visit (Visit 1) and/or 1st vaccination visit (Visit 2) will not be eligible for participation in this study. All Investigator assessment-based judgments must be carefully and fully documented in the source documents:

  1. According to the Investigator's opinion, significant acute or chronic, uncontrolled medical or neuropsychiatric illness.

Acute disease is defined as presence of any moderate or severe acute illness with or without a fever within 48 hours prior to the Screening visit (Visit 1) and/or 1st vaccination visit (Visit 2).

'Uncontrolled' is defined as:

* Requiring a new medical or surgical treatment during the three months prior to study vaccine administration;
* Requiring any significant change in a chronic medication (i.e. drug, dose, frequency) during the three months prior to study vaccine administration due to uncontrolled symptoms or drug toxicity unless the innocuous nature of the medication change meets the criteria outlined in inclusion criterion no. 8 and is appropriately justified by the Investigator.

Investigator discretion is permitted with this exclusion criterion. 2. Any confirmed or suspected current immunosuppressive condition or immunodeficiency, including cancer, HIV, hepatitis B or C infection (subjects with a history of cured hepatitis B or C infection without any signs of immunodeficiency at present time are allowed). Investigator discretion is permitted with this exclusion criterion; 3. Current autoimmune disease (such as rheumatoid arthritis, systemic lupus erythematosus or multiple sclerosis). Investigator discretion is permitted with this exclusion criterion. Subjects may be eligible to participate with appropriate written justification in the source document. For example, subjects with a history of autoimmune disease who are disease-free without treatment for three years or more, subjects receiving stable thyroid replacement therapy, and subjects with mild psoriasis (i.e. a small number of minor plaques requiring no systemic treatment) are eligible for participation; 4. Administration of any medication or treatment that may alter the vaccine immune responses, such as:

* Systemic glucocorticoids at a dose exceeding 10 mg of prednisone (or equivalent) per day for more than seven consecutive days or for 10 or more days in total, within one month prior to the 1st vaccination visit (Visit 2). Inhaled, nasal, ophthalmic, dermatological, and other topical glucocorticoids are permitted;
* Cytotoxic, antineoplastic, or immunosuppressant drugs - within 36 months prior to 1st vaccination visit (Visit 2);
* Any immunoglobulin preparations, blood products, or blood transfusion - within 6 months prior to 1st vaccination visit (Visit 2); 5. Administration of any vaccine within 14 days prior to 1st vaccination visit (Visit 2); planned administration of any vaccine during the study (up to Day 28). Immunization on an emergency basis during the study will be evaluated on case-by-case basis by the Investigator; 6. Administration of any other SARS-CoV-2/COVID-19 vaccine, or other experimental coronavirus vaccine at any time prior to or during the study; 7. At screening (Visit 1), subjects found to be seropositive for prior SARS-COV-2 infection based on N-protein ELISA or positive for SARS-COV-2 PCR test; 8. Subjects with previous diagnosis of COVID-19 or previous positive SARS-CoV-2 infection 9. Use of any investigational or non-registered product within 30 days or 5 half-lives, whichever is longer, prior to 1st vaccination visit (Visit 2), or planned use during the study period. Subjects who are in a prolonged post-administration observation period of another investigational or marketed drug clinical study, for which there is no ongoing exposure to the investigational or marketed product and all scheduled on-site visits are completed, will be allowed to take part in this study, if all other eligibility criteria are met; 10. Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at injection site that may interfere with injection site reaction rating. Investigator discretion is permitted with this exclusion criterion: 11. Use of any prescription antiviral drugs with the intention of COVID-19 prophylaxis, including those that are thought to be effective for prevention of COVID-19 but have not been licensed for this indication, within one month prior to 1st vaccination visit (Visit 2); 12. Use of prophylactic medications (e.g. antihistamines [H1 receptor antagonists], nonsteroidal anti-inflammatory drugs [NSAIDs], systemic and topical glucocorticoids, non-opioid and opioid analgesics) within 24 hours prior to the 1st vaccination (Visit 2) to prevent or pre-empt symptoms due to vaccination; 13. History of a serious allergic response to any of the constituents of MT-2766; 14. History of a documented anaphylactic reactions to plants or plant components (including tobacco, fruits, and nuts); 15. Personal or family (first-degree relatives) history of narcolepsy; 16. Subjects with a history of Guillain-Barré Syndrome; 17. Any female subject who has a definitely or possibly positive pregnancy test result prior to vaccination or who is lactating; 18. As a result of the medical screening process, the Investigator considers the subject not suitable for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2023-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Medicago
Locations (3):
- Japan (3):
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Low dose arm is open-label, not randomized arm and was not enrolled. It was described in the protocol that the study may be completed even if fewer than planned number of subjects in Low dose arm are enrolled.
Groups:
- MT-2766 High Dose (3.75 µg): Subjects received two doses of MT-2766 high dose (3.75 µg) given 21 days apart into the deltoid region of the alternating arm (each arm will be injected once).
- Placebo: Subjects received two doses of placebo given 21 days apart into the deltoid region of the alternating arm (each arm will be injected once).
Period: Up to Day 42
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Started | 102 | 26
Completed | 100 | 26
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: After Day 43
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Started | 100 | 26
Completed | 0 | 0
Not Completed | 100 | 26
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Public vaccination | 6 | 8
Not completed — Difficult to go to the hospital due to moving | 1 | 0
Not completed — Study Terminated by Sponsor | 88 | 16

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized subjects who received at least 1 dose of the investigational product.
  After randomization, one subject withdrew before receiving investigational product at the subject's request.
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo | Total
Number analyzed (Participants) | 101 | 26 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 25 | 122
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (11.3) | 46.8 (11.9) | 46.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 15 | 51
  Male | 65 | 11 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 101 | 26 | 127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 101 | 26 | 127
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Immediate Adverse Events (AEs) According to Severity, and Investigator-assessed Causality
Description: Immediate AEs are defined as any solicited AEs and unsolicited AEs occurring within 30 minutes after vaccination. The causal relationship of all solicited AEs to investigational product was analyzed as related.
Time Frame: Within 30 minutes after each vaccination
Population: Safety population included all randomized subjects who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 101 | 26
percentage of participants
  Percentage of Participants with Immediate Solicited AEs | 11.9 | 7.7
  Severity of Immediate Solicited AE: Mild | 11.9 | 7.7
  Severity of Immediate Solicited AE: Moderate | 0 | 0
  Severity of Immediate Solicited AE: Severe | 0 | 0
  Severity of Immediate Solicited AE: Potentially life-threatening | 0 | 0
  Percentage of Participants with Immediate Unsolicited AE | 1.0 | 0
  Severity of Immediate Unsolicited AE: Mild | 1.0 | 0
  Severity of Immediate Unsolicited AE: Moderate | 0 | 0
  Severity of Immediate Unsolicited AE: Severe | 0 | 0
  Severity of Immediate Unsolicited AE: Potentially life-threatening | 0 | 0
  Percentage of Participants with Immediate Related Unsolicited AE | 1.0 | 0

2. Primary Outcome: Percentage of Participants With Solicited AEs According to Severity
Description: Solicited AEs are defined the following; (i) local AEs (injection site erythema, injection site swelling, injection site induration, and injection site pain) and (ii) systemic AEs (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck)．
Time Frame: Within 7 days after each vaccination
Population: Safety population included all randomized subjects who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 101 | 26
percentage of participants
  Percentage of Participants with Solicited AE | 91.1 | 42.3
  Severity of Solicited AE: Mild | 60.4 | 38.5
  Severity of Solicited AE: Moderate | 24.8 | 3.8
  Severity of Solicited AE: Severe | 5.0 | 0
  Severity of Solicited AE: Potentially life-threatening | 0 | 0
  Percentage of Participants with Solicited Local AE | 85.1 | 11.5
  Severity of Solicited Local AE: Mild | 76.2 | 11.5
  Severity of Solicited Local AE: Moderate | 6.9 | 0
  Severity of Solicited Local AE: Severe | 2.0 | 0
  Severity of Solicited Local AE: Potentially life-threatening | 0 | 0
  Percentage of Participants with Solicited Systemic AE | 70.3 | 38.5
  Severity of Solicited Systemic AE: Mild | 45.5 | 34.6
  Severity of Solicited Systemic AE: Moderate | 20.8 | 3.8
  Severity of Solicited Systemic AE: Severe | 3.0 | 0
  Severity of Solicited Systemic AE: Potentially life-threatening | 0 | 0

3. Primary Outcome: Percentage of Participants With Unsolicited AEs According to Severity, and Investigator-assessed Causality
Time Frame: Within 21 days after each vaccination
Population: Safety population included all randomized subjects who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 101 | 26
percentage of participants
  Percentage of Participants with Unsolicited AEs | 18.8 | 26.9
  Severity of Unsolicited AE: Mild | 15.8 | 26.9
  Severity of Unsolicited AE: Moderate | 3.0 | 0
  Severity of Unsolicited AE: Severe | 0.0 | 0
  Severity of Unsolicited AE: Potentially life-threatening | 0 | 0
  Percentage of Participants with Related Unsolicited AE | 12.9 | 0

4. Primary Outcome: Percentage of Participants With Serious AEs (SAEs), Medically Attended AEs (MAAEs), AEs Leading to Withdrawal, AEs of Special Interest (AESIs), and Deaths
Description: AESIs include vaccine-associated enhanced diseases, hypersensitivity reactions, and potential immune-mediated diseases
Time Frame: Within 21 days after each vaccination
Population: Safety population included all randomized subjects who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 101 | 26
percentage of participants
  Percentage of Participants with SAEs | 0 | 0
  Percentage of Participants with MAAEs | 3.0 | 11.5
  Percentage of Participants with AEs Leading to Study Withdrawal | 0 | 0
  Percentage of Participants with AESIs | 2.0 | 0
  Percentage of Participants with Deaths | 0 | 0

5. Primary Outcome: SARS-CoV-2 Neutralizing Antibody (Nab) Responses: GMT
Description: Geometric mean neutralizing antibody titer (GMT)
Time Frame: Day 0 (before 1st vaccination), Day 21 (21 days after 1st vaccination and before 2nd vaccination), and Day 42 (21 days after 2nd vaccination)
Population: Immunogenicity Per Protocol population included all randomized subjects who do not have any major protocol violations, and who received the investigational product. For the Day 21 analysis, this included the subjects who received the first vaccine dose and had Day 0 and Day 21 immunogenicity sample collections. For the Day 42 analysis, this included the subjects who received both vaccine doses and had Day 0 and Day 42 immunogenicity sample collections.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 99 | 26
titer
  GMT: Day 0 | 6.6 [5.5 to 8.0] | 6.9 [4.5 to 10.6]
  GMT: Day 21: number analyzed (Participants) | 95 | 25
  GMT: Day 21 | 43.9 [31.9 to 60.3] | 7.0 [4.3 to 11.5]
  GMT: Day 42: number analyzed (Participants) | 97 | 25
  GMT: Day 42 | 912.6 [733.6 to 1135.1] | 7.0 [4.5 to 11.0]

6. Primary Outcome: SARS-CoV-2 Neutralizing Antibody (Nab) Responses: GMFR
Description: Geometric mean fold rise (GMFR) is defined as the ratio of geometric mean antibody titer (GMT) based on that of Day 0 (i.e. Day 21/Day 0 and Day 42/Day 0).
Time Frame: Day 21 (21 days after 1st vaccination and before 2nd vaccination), and Day 42 (21 days after 2nd vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 99 | 26
fold rise
  GMFR: Day 21/Day 0: number analyzed (Participants) | 95 | 25
  GMFR: Day 21/Day 0 | 6.55 [5.20 to 8.26] | 1.03 [0.66 to 1.62]
  GMFR: Day 42/Day 0: number analyzed (Participants) | 97 | 25
  GMFR: Day 42/Day 0 | 136.75 [112.15 to 166.74] | 1.04 [0.71 to 1.54]

7. Primary Outcome: SARS-CoV-2 Neutralizing Antibody (Nab) Responses
Description: Seroconversion (SC) rate. SC rate is defined as the proportion of subjects achieving SC in the analysis set i.e. subjects with:
  * For subjects with detectable Nab titer at Day 0 (i.e. baseline Nab titer ≥10): a ≥ 4-fold increase in Nab titers between Day 0 and Day 21/42, respectively.
  * For subjects with undetectable Nab titer at Day 0 (i.e. baseline Nab titer < 10): Nab titer of ≥ 40 on Day 21/42, respectively.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SC
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 99 | 26
percentage of subjects achieving SC
  Day 21: number analyzed (Participants) | 95 | 25
  Day 21 | 38.9 [29.1 to 49.5] | 0 [0.0 to 13.7]
  Day 42: number analyzed (Participants) | 97 | 25
  Day 42 | 99.0 [94.4 to 100.0] | 0 [0.0 to 13.7]

8. Primary Outcome: SARS-CoV-2-specific T Helper 1 (Th1) Cell-mediated Immune (CMI) Responses
Description: Using the interferon-γ enzyme-linked immunospot (ELISpot) assay. Unit of Measure: Spot-Forming Cell (SFC)/10^6 Peripheral Blood Mononuclear Cells (PBMC)
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: SFC/10^6 PBMC
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 99 | 26
SFC/10^6 PBMC
  Day 0: number analyzed (Participants) | 80 | 22
  Day 0 | 188.0 [73.0 to 258.0] | 277.5 [120.0 to 450.0]
  Day 21: number analyzed (Participants) | 85 | 24
  Day 21 | 265.5 [128.0 to 635.0] | 330.0 [233.0 to 465.0]
  Day 42: number analyzed (Participants) | 95 | 21
  Day 42 | 1173.0 [1010.0 to 1305.0] | 413.0 [43.0 to 835.0]

9. Primary Outcome: SARS-CoV-2-specific T Helper 2 (Th2) CMI Responses
Description: Using the interleukin-4 ELISpot assay
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: SFC/10^6 PBMC
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 99 | 26
SFC/10^6 PBMC
  Day 0: number analyzed (Participants) | 92 | 24
  Day 0 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Day 21: number analyzed (Participants) | 90 | 26
  Day 21 | 0.0 [0.0 to 75.0] | 0.0 [0.0 to 0.0]
  Day 42: number analyzed (Participants) | 91 | 25
  Day 42 | 619.0 [540.0 to 786.0] | 0.0 [0.0 to 0.0]

10. Secondary Outcome: Percentage of Participants With Serious AEs (SAEs), Medically Attended AEs (MAAEs), AEs Leading to Withdrawal, AEs of Special Interest (AESIs), and Deaths
Description: AESIs include vaccine-associated enhanced diseases, hypersensitivity reactions, and potential immune-mediated diseases.
Time Frame: Day 0 (after 1st vaccination) to end of study, on average the study duration by the termination is 334 days.
Population: Safety population included all randomized subjects who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 101 | 26
percentage of participants
  Percentage of Participants with SAEs | 2.0 | 7.7
  Percentage of Participants with MAAEs | 31.7 | 46.2
  Percentage of Participants with AEs Leading to Study Withdrawal | 0 | 0
  Percentage of Participants with AESIs | 2.0 | 0
  Percentage of Participants with Deaths | 0 | 0

11. Secondary Outcome: SARS-CoV-2 Neutralizing Antibody (Nab) Responses: GMT
Description: Geometric mean neutralizing antibody titer (GMT)
Time Frame: Day 128 and Day 201
Population: This analysis population included randomized subjects who had no major protocol violations and received investigational drug (MT-2766 n=100, Placebo n=26). For the Day 128, analysis included the subjects who received both doses and had Day 0 and 128 sample collections (MT-2766 n=94, Placebo n=25). For the Day 201, analysis included the subjects who received both doses and had Day 0 and 201 sample collections (MT-2766 n=90, Placebo n=22).
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 94 | 25
titer
  GMT: Day 128 | 196.5 [147.0 to 262.7] | 8.5 [4.6 to 15.8]
  GMT: Day 201: number analyzed (Participants) | 90 | 22
  GMT: Day 201 | 139.9 [99.5 to 196.8] | 8.3 [4.2 to 16.4]

12. Secondary Outcome: SARS-CoV-2 Neutralizing Antibody (Nab) Responses: GMFR
Description: Geometric mean fold rise (GMFR)
Time Frame: Day 128 and Day 201
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 94 | 25
fold rise
  GMFR: Day 128/Day 0 | 29.17 [22.60 to 37.65] | 1.22 [0.74 to 2.00]
  GMFR: Day 201/Day 0: number analyzed (Participants) | 90 | 22
  GMFR: Day 201/Day 0 | 22.63 [16.55 to 30.94] | 1.17 [0.62 to 2.21]

13. Secondary Outcome: Seroconversion (SC) Rate of SARS-CoV-2 Neutralizing Antibody
Description: SC rate is defined as the proportion of subjects achieving SC in the analysis set i.e. subjects with:
  * For subjects with detectable Nab titer at Day 0 (i.e. baseline Nab titer ≥10): a ≥ 4-fold increase in Nab titers between Day 0 and Day 128/201, respectively.
  * For subjects with undetectable Nab titer at Day 0 (i.e. baseline Nab titer < 10): Nab titer of ≥ 40 on Day 128/201, respectively.
Time Frame: Day 128 and Day 201
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ％
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 94 | 25
％
  SC rate: Day 128 | 90.4 [82.6 to 95.5] | 4.0 [0.1 to 20.4]
  SC rate: Day 201: number analyzed (Participants) | 90 | 22
  SC rate: Day 201 | 77.8 [67.8 to 85.9] | 4.5 [0.1 to 22.8]

14. Secondary Outcome: SARS-CoV-2-specific T Helper 1 (Th1) Cell-mediated Immune (CMI) Responses
Description: Using the interferon-γ enzyme-linked immunospot (ELISpot) assay.
Time Frame: Days 201
Population: Immunogenicity Per Protocol population included all randomized subjects who do not have any major protocol violations, and who received the investigational product. For the Day 128 analysis, this should include the subjects who received both vaccine doses and had Day 0 and Day 128 immunogenicity sample collections. For the Day 201 analysis, this should include the subjects who received both vaccine doses and had Day 0 and Day 201 immunogenicity sample collections.
Measure: Median (95% Confidence Interval); unit: SFC/10^6 PBMC
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 85 | 18
SFC/10^6 PBMC | 948.0 [815.0 to 1103.0] | 171.50 [0.00 to 295.00]

15. Secondary Outcome: SARS-CoV-2-specific T Helper 2 (Th2) CMI Responses
Description: Using the interleukin-4 ELISpot assay
Time Frame: Days 201
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: SFC/10^6 PBMC
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 87 | 19
SFC/10^6 PBMC | 375.0 [302.0 to 516.0] | 0.0 [0.0 to 0.0]

16. Secondary Outcome: SARS-CoV-2-specific Antibody Responses (Total IgG): GMT
Description: Geometric mean neutralizing antibody titer (GMT)
Time Frame: Day 0，Day 21，Day 42，Day 128 and Day 201
Population: This analysis population included randomized subjects who had no major protocol violations and received investigational drug (MT-2766 n=100, Placebo n=26). For the Day 21, analysis included the subjects who received the 1st dose and had Day 0 and 21 sample collections. For the Day 42, 128, and 201, analyses included the subjects who received two doses and had Day 0 and the each time point sample collections. See the table below for the number of analyzed subjects at each time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 100 | 26
titer
  GMT: Day 0 | 103.6 [72.8 to 147.6] | 119.5 [52.5 to 271.7]
  GMT: Day 21: number analyzed (Participants) | 98 | 26
  GMT: Day 21 | 2258.3 [1529.5 to 3334.3] | 118.6 [52.1 to 270.0]
  GMT: Day 42: number analyzed (Participants) | 97 | 25
  GMT: Day 42 | 95159.8 [78038.0 to 116038.2] | 114.3 [50.6 to 257.9]
  GMT: Day 128: number analyzed (Participants) | 94 | 26
  GMT: Day 128 | 24391.9 [17875.1 to 33284.5] | 147.0 [59.4 to 363.7]
  GMT: Day 201: number analyzed (Participants) | 90 | 22
  GMT: Day 201 | 15429.0 [10934.6 to 21770.8] | 216.6 [80.2 to 584.7]

17. Secondary Outcome: SARS-CoV-2-specific Antibody Responses (Total IgG): GMFR
Description: Geometric mean fold rise (GMFR)
Time Frame: Day 0，Day 21，Day 42，Day 128 and Day 201
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 98 | 26
fold rise
  GMFR: Day 21/Day 0 | 22.34 [16.94 to 29.47] | 1.02 [0.60 to 1.75]
  GMFR: Day 42/Day 0: number analyzed (Participants) | 97 | 25
  GMFR: Day 42/Day 0 | 917.37 [738.51 to 1139.54] | 1.03 [0.67 to 1.57]
  GMFR: Day 128/Day 0: number analyzed (Participants) | 94 | 26
  GMFR: Day 128/Day 0 | 245.38 [181.54 to 331.67] | 1.34 [0.75 to 2.38]
  GMFR: Day 201/Day 0: number analyzed (Participants) | 90 | 22
  GMFR: Day 201/Day 0 | 176.32 [125.47 to 247.77] | 1.95 [0.98 to 3.90]

18. Secondary Outcome: Seroconversion (SC) Rate of SARS-CoV-2-specific Antibody Responses (Total IgG):
Description: SC rate is defined as the proportion of subjects achieving SC in the analysis set i.e. subjects with:
  * For subjects with detectable Nab titer at Day 0 (i.e. baseline Nab titer ≥10): a ≥ 4-fold increase in Nab titers between Day 0 and Day 21/42/128/201, respectively.
  * For subjects with undetectable Nab titer at Day 0 (i.e. baseline Nab titer < 10): Nab titer of ≥ 40 on Day 21/42, respectively.
Time Frame: Day 0，Day 21，Day 42，Day 128 and Day 201
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SC
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
Number analyzed (Participants) | 98 | 26
percentage of subjects achieving SC
  SC rate: Day 21 | 83.7 [74.8 to 90.4] | 0.0 [0.0 to 13.2]
  SC rate: Day 42: number analyzed (Participants) | 97 | 25
  SC rate: Day 42 | 97.9 [92.7 to 99.7] | 0.0 [0.0 to 13.7]
  SC rate: Day 128: number analyzed (Participants) | 94 | 26
  SC rate: Day 128 | 96.8 [91.0 to 99.3] | 11.5 [2.4 to 30.2]
  SC rate: Day 201: number analyzed (Participants) | 90 | 22
  SC rate: Day 201 | 95.6 [89.0 to 98.8] | 18.2 [5.2 to 40.3]

ADVERSE EVENTS:
Time Frame: Day 0 (after 1st vaccination) to end of study, on average the study duration by the termination is 334 days.
Description: Data were collected based on regular investigator assessment and laboratory testing, self-reporting by participants and subject diary. For solicited AEs, prespecified AEs were collected up to 7 days after each administration using the subject diary.
Arm/Group | MT-2766 High Dose (3.75 µg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/101 | 2/26
Other Adverse Events (participants affected / at risk) | 92/101 | 11/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-2766 High Dose (3.75 µg) (N=101) | Placebo (N=26)
COVID-19 (Infections and infestations) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-2766 High Dose (3.75 µg) (N=101) | Placebo (N=26)
Induration (General disorders) | 36 | 0
Pain (General disorders) | 84 | 3
Redness (Skin and subcutaneous tissue disorders) | 12 | 0
Chills (General disorders) | 44 | 1
Fatigue (General disorders) | 50 | 6
Feeling of General Discomfort (General disorders) | 39 | 5
Feeling of Swelling in the Neck (General disorders) | 9 | 1
Fever (General disorders) | 15 | 0
Headache (Nervous system disorders) | 47 | 5
Joint Aches (Musculoskeletal and connective tissue disorders) | 28 | 1
Muscle Aches (Musculoskeletal and connective tissue disorders) | 44 | 0
Swelling (General disorders) | 30 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT05065619/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT05065619/SAP_002.pdf